CLINICAL TRIAL: NCT01808651
Title: A Phase 3, Open-label, Long-Term Study to Evaluate the Safety of LY110140 Once Daily Dosing for 52-week in Japanese Patients With Major Depressive Disorder
Brief Title: A Study of Fluoxetine in Major Depressive Disorder (MDD) Long-Term Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14596; B1Y-JE-HCLW (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine (Experimental): Flexible dosing of 20 to 40 milligrams (mg) administered orally, once daily, for approximately 52 weeks
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Administered orally
  Other Names: LY110140; Fluoxetine Hydrochloride; Prozac; Sarafem

SUMMARY:
This study will evaluate the safety and effectiveness of fluoxetine flexible dosing in the treatment of MDD in adult Japanese participants.

Participants who complete the short-term treatment phase of Study B1Y-JE-HCLV (NCT#: NCT01808612) will be allowed to enroll in this study, and receive fluoxetine treatment for an additional 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have completed Study B1Y-JE-HCLV (NCT#:NCT01808612)
* Agree to abstain from sexual activity or to use a reliable method of birth control

Exclusion Criteria:

* Significant suicidal risk
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, or post-traumatic stress disorder
* Have a history of substance abuse or dependence within the past 6 months, excluding caffeine and nicotine
* Need to use thioridazine or pimozide during the study
* Have a positive urine drug screen for drugs with abuse potential
* Female participants who are either pregnant, nursing, or have recently given birth, or male participants who are planning for their partners to be or become pregnant
* Have frequent or severe allergic reactions to multiple medications
* Have a serious or unstable medical illness or condition, or psychological condition
* Participants deemed ineligible by the investigator or sub-investigator for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 2 study periods for Japanese participants who completed acute treatment in Study B1Y-JE-HCLV(NCT#: NCT01808612): Study period I was a 52-week open-label treatment period with fluoxetine 20 to 40 milligrams (mg), administered once daily, and Study period II was a 2-wk observation phase following discontinuation of fluoxetine.
Groups:
- PLA/FLX: Period 1: Participants (Pts) randomized to placebo in Study B1Y-JE-HCLV transitioned to fluoxetine 20 to 40 mg capsules administered orally, once daily, for 52 weeks in Study B1Y-JE-HCLW.
  Period 2: 2-week observation phase following discontinuation (DC'd) of fluoxetine.
- FLX20/FLX: Period 1: Participants randomized to fluoxetine 20 mg /day in Study B1Y-JE-HCLV and continued on fluoxetine 20 to 40 mg capsules administered orally, once daily, for 52 weeks in Study B1Y-JE-HCLW.
  Period 2: 2-week observation phase following discontinuation of fluoxetine.
- FLX40/FLX: Period 1: Participants randomized to fluoxetine 40 mg/day in Study B1Y-JE-HCLV and continued on fluoxetine 20 to 40 mg capsules administered orally, once daily, for 52 weeks in Study B1Y-JE-HCLW.
  Period 2: 2-week observation phase following discontinuation of fluoxetine.
Period: Study Period 1
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Started | 99 | 65 | 36
Received at Least One Dose of Study Drug | 98 | 65 | 36
Completed | 73 | 48 | 31
Not Completed | 26 | 17 | 5
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Physician Decision | 3 | 2 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Adverse Event | 10 | 4 | 1
Not completed — Participant Decision | 9 | 7 | 3
Period: Study Period 2
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Started | 77 | 52 | 33
Completed | 77 (9 Pts who DC'd from Study Period 1 and 68 Pts who completed Study Period 1 entered Study Period 2.) | 52 (5 Pts who DC'd from Study Period 1 and 47 Pts who completed Study Period 1 entered Study Period 2.) | 33 (3 Pts who DC'd from Study Period 1 and 30 pts who completed Study Period 1 entered Study Period 2.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PLA/FLX (Placebo/Fluoxetine): Participants randomized to placebo in Study B1Y-JE-HCLV and transitioned to fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- FLX20/FLX: Participants randomized to fluoxetine 20 mg/day in Study B1Y-JE-HCLV and continued on fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- FLX40/FLX: Participants randomized to fluoxetine 40 mg/day in Study B1Y-JE-HCLV and continued on fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- Total: Total of all reporting groups
Arm/Group | PLA/FLX (Placebo/Fluoxetine) | FLX20/FLX | FLX40/FLX | Total
Number analyzed (Participants) | 98 | 65 | 36 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.60 (12.95) | 39.72 (10.91) | 41.20 (10.51) | 39.44 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 33 | 19 | 99
  Male | 51 | 32 | 17 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 98 | 65 | 36 | 199
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 98 | 65 | 36 | 199

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) or Serious AEs (SAEs)
Time Frame: Baseline through Week 52.
Population: Participants who received at least 1 dose of the study drug were evaluated for AEs and SAEs. SAE reported for 1 participant (FLX20/FLX) was a pre-existing condition prior to Study Period 1 that became an SAE after Study Period 1.
Measure: Number; unit: participants
Groups:
- PLA/FLX: Participants randomized to placebo in Study B1Y-JE-HCLV and transitioned to fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 65 | 36
participants
  Participants with >=1 SAE | 2 | 1 | 0
  Participants with >=1 AEs | 75 | 46 | 29

2. Primary Outcome: Number of Participants With Suicidal Behaviors and Ideations Collected by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline through Week 52
Population: Participants who received at least 1 dose of study drug with at least 1 post-baseline C-SSRS score during Study Period 1.
Measure: Number; unit: participants
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 65 | 36
participants | 8 | 4 | 0

3. Secondary Outcome: Mean Change From Baseline to Week 52 on the 21-Item Hamilton Depression Rating Scale (HAMD21) Total Score
Description: HAMD21 is a 21-item assessment used to measure depression severity. Items were rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score ranging from 0 (not at all depressed) to 64 (severely depressed). Least squares (LS) means were calculated using mixed-model repeated measures (MMRM) adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline HAMD21 total score.
Time Frame: Baseline, Week 52
Population: Participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 total score during Study Period 1.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 64 | 36
units on a scale | -10.04 (0.73) | -11.25 (0.90) | -11.70 (1.16)

4. Secondary Outcome: Percentage of Participants Achieving a Response at Week 52
Description: The percentage of participants achieving a response (defined as a ≥50% improvement from baseline on the HAMD21 total score) was calculated by dividing the number of participants achieving a response at last observation by the total number of participants at risk, multiplied by 100.
Time Frame: Baseline, up to Week 52
Population: Participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 total score during the Treatment Period. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: Percentage of participants
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 65 | 36
Percentage of participants | 68 | 65 | 83

5. Secondary Outcome: Percentage of Participants Achieving a Remission at Week 52
Description: The percentage of participants achieving a remission (defined as a HAMD21 total score ≤7) was calculated by dividing the number of participants achieving a remission at last observation by the total number of participants at risk, multiplied by 100.
Time Frame: up to Week 52
Population: Participants who received at least 1 dose of study drug with a baseline (which had not achieved remission threshold criteria) and had at least 1 post-baseline HAMD21 total score during the Treatment Period. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 86 | 60 | 33
percentage of participants | 64 | 57 | 76

6. Secondary Outcome: Mean Change From Baseline to Week 52 on the Clinical Global Impression of Severity (CGI-S) Scale
Description: CGI-S measures severity of illness at the time of assessment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). LS means were calculated using MMRM adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline CGI-S score.
Time Frame: Baseline, Week 52
Population: Participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline CGI-S score during the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 64 | 36
units on a scale | -1.41 (0.10) | -1.45 (0.13) | -1.64 (0.16)

7. Secondary Outcome: Mean Change From Baseline to Week 52 on the HAMD21 Subscale Scores
Description: HAMD17 total scores and subscale scores from the HAMD21 are presented. HAMD17 is a 17-item assessment of depression severity (total scores range from 0-52). The Maier subscale (Items 1, 2, 7-10) represents the core symptoms of depression (0-24). Anxiety/Somatization subscale (Items 10-13, 15, 17) evaluates severity of psychic and somatic manifestations of anxiety as well as agitation (0-18). Retardation/Somatization subscale (Items 1, 7, 8, 14) evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation (0-14). Sleep subscale (Items 4-6) assesses insomnia (0-6). Individual item scores may range from 0-4 or 0-2. Higher scores indicate more severe symptoms. LS means were calculated using MMRM adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline score.
Time Frame: Baseline, Week 52
Population: Participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 subscale score. LSM (least square mean) and SE (standard error) are from visit 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 64 | 36
units on a scale
  HAMD17 total scale | -9.06 (0.67) | -10.20 (0.83) | -10.51 (1.07)
  Maier subscale score | -4.73 (0.37) | -5.55 (0.46) | -5.02 (0.60)
  Anxiety/Somatization subscale score | -3.08 (0.25) | -3.16 (0.31) | -3.61 (0.39)
  Retardation/Somatization subscale score | -3.45 (0.26) | -3.98 (0.32) | -3.55 (0.42)
  Sleep subscale score | -1.49 (0.15) | -1.34 (0.18) | -1.95 (0.23)

8. Secondary Outcome: Change From Baseline to Week 52 in Sheehan Disability Scale (SDS) Total Score and Subscale Scores
Description: SDS was completed by the participant and was used to assess the effect of the participant's symptoms on their work/school (Item 1), social life/leisure activities (Item 2), and family life/home responsibilities (Item 3). Each item was measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total score was the sum of the 3 items and ranged from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. LS means were calculated using analysis of covariance (ANCOVA) adjusting for treatment, pooled investigative site, and baseline SDS score.
Time Frame: Baseline up to 52 weeks
Population: Participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline SDS score. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PLA/FLX | FLX20/FLX | FLX40/FLX
Number analyzed (Participants) | 98 | 64 | 36
units on a scale
  SDS Total Score | -6.53 (0.78) | -6.17 (0.97) | -6.14 (1.28)
  Work/School subscale (N:85, 60, 28) | -2.46 (0.32) | -2.62 (0.38) | -2.24 (0.56)
  Social/Leisure subscale (N:98, 64, 36) | -2.11 (0.28) | -2.11 (0.35) | -2.06 (0.47)
  Family/Home subscale (N:98,64,36) | -1.93 (0.25) | -1.55 (0.31) | -2.01 (0.41)

ADVERSE EVENTS:
Description: SAE "Asthma" reported for 1 participant (FLX20/FLX) was a pre-existing condition prior to Study Period 1 that became an SAE after Study Period 2; however, SAE "Asthma" was reported in both Study Period 1 and Study Period 2 for this participant.
Groups:
- Study Period 1 PLA/FLX: Participants randomized to placebo in Study B1Y-JE-HCLV and transitioned to fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- Study Period 1 FLX20/FLX: Participants randomized to fluoxetine 20 mg/day in Study B1Y-JE-HCLV and continued on fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- Study Period 1 FLX40/FLX: Participants randomized to fluoxetine 40 mg/day in Study B1Y-JE-HCLV and continued on fluoxetine (20-40 mg/day) in Study B1Y-JE-HCLW.
- Study Period 2 Discontinued From PLA/FLX: Participants in the PLA/FLX group in Study Period 1, and discontinuing from fluoxetine in Study Period 2,
- Study Period 2 Discontinued From FLX20/FLX: Participants in the FLX20/FLX group in Study Period 1, and discontinuing from fluoxetine in Study Period 2.
- Study Period 2 Discontinued From FLX40/FLX: Participants in the FLX40/FLX group in Study Period 1, and discontinuing from fluoxetine in Study Period 2.
Arm/Group | Study Period 1 PLA/FLX | Study Period 1 FLX20/FLX | Study Period 1 FLX40/FLX | Study Period 2 Discontinued From PLA/FLX | Study Period 2 Discontinued From FLX20/FLX | Study Period 2 Discontinued From FLX40/FLX
Serious Adverse Events (participants affected / at risk) | 2/98 | 1/65 | 0/36 | 0/77 | 1/52 | 0/33
Other Adverse Events (participants affected / at risk) | 74/98 | 46/65 | 29/36 | 5/77 | 7/52 | 1/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Period 1 PLA/FLX (N=98) | Study Period 1 FLX20/FLX (N=65) | Study Period 1 FLX40/FLX (N=36) | Study Period 2 Discontinued From PLA/FLX (N=77) | Study Period 2 Discontinued From FLX20/FLX (N=52) | Study Period 2 Discontinued From FLX40/FLX (N=33)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Period 1 PLA/FLX (N=98) | Study Period 1 FLX20/FLX (N=65) | Study Period 1 FLX40/FLX (N=36) | Study Period 2 Discontinued From PLA/FLX (N=77) | Study Period 2 Discontinued From FLX20/FLX (N=52) | Study Period 2 Discontinued From FLX40/FLX (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 32 (43) | 20 (27) | 15 (26) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/47 (0) | 1/33 (1) | 0/19 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/47 (0) | 1/33 (1) | 0/19 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 6 (9) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7) | 5 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Activation syndrome (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichotillomania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/47 (1) | 1/33 (7) | 1/19 (1) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1/47 (1) | 0/33 (0) | 0/19 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days